CLINICAL TRIAL: NCT03783936
Title: A Single Arm, Multi-center Phase 2 Trial of mFOLFOX6 + Trastuzumab + Avelumab in First-line, Metastatic, HER2-amplified Gastric and Esophageal Adenocarcinomas
Brief Title: Trial of mFOLFOX6 + Trastuzumab + Avelumab in Gastric and Esophageal Adenocarcinomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ashwin Somasundaram (Other)
Collaborators: EMD Serono (Industry); University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor-Investigator, Ashwin Somasundaram, Sponsor-Investigator, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCRN GI17-319
Record Dates: First submitted 2018-12-19; First posted 2018-12-21 (Actual); Results first posted 2023-12-19 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-11

CONDITIONS: Gastric Adenocarcinoma; Esophageal Adenocarcinoma; Metastasis; HER-2 Gene Amplification
MeSH Terms: conditions — Adenocarcinoma Of Esophagus; Neoplasm Metastasis | interventions — Oxaliplatin; Leucovorin; Fluorouracil; Trastuzumab; avelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Induction and Maintenance (Other): Cycles 1-9; Induction; Cycle = 14 days
  mFOLFOX6
  * oxaliplatin 85 mg/m2 IV Day 1 and
  * leucovorin 400 mg/m2 IV Day 1 and
  * 5 fluorouracil 400 mg/m2 IV bolus and 2400 mg/m2 IV over 46 hours Day 1 and
  Trastuzumab 6 mg/kg IV loading dose C1D1 then Trastuzumab 4 mg/kg IV Day 1 and
  Avelumab 800 mg IV Day 1
  Cycles 10 and subsequent; Maintenance; Cycle = 14 days
  Trastuzumab 4 mg/kg Day 1 and Avelumab 800 mg Day 1
  Interventions: Drug: Oxaliplatin; Drug: Leucovorin; Drug: 5 fluorouracil; Drug: Trastuzumab; Drug: Avelumab

INTERVENTIONS:
Drug: Oxaliplatin — Oxaliplatin 85 mg/m2
Drug: Leucovorin — Leucovorin 400 mg/m2
Drug: 5 fluorouracil — 5 fluorouracil 400 mg/m2 bolus and 2400 mg/m2 continuous infusion
Drug: Trastuzumab — Trastuzumab 6 mg/kg loading dose C1D1 then 4 mg/kg Day 1
Drug: Avelumab — Avelumab 800 mg

SUMMARY:
The initial intent of the study was to be a multi-center single-arm open-label Simon's two-stage Phase II clinical trial of first-line mFOLFOX6 + trastuzumab + avelumab in metastatic HER2-amplified gastric and esophageal adenocarcinomas.

Accrual will halt after completion of Stage I (enrollment of 18 patients). This decision is not due to safety issues. Subjects currently on treatment will continue until criteria as defined in the protocol is met.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent and HIPAA authorization for release of personal health information prior to registration.
2. Age ≥ 18 years at the time of consent.
3. ECOG Performance Status of 0 or 1.
4. Histologically confirmed esophageal, gastroesophageal junction, or gastric adenocarcinoma, with unresectable or metastatic disease documented on diagnostic imaging studies.
5. HER2 amplification confirmed by standard of care testing of tumor specimen (3+ by immunohistochemistry, or 2+ on IHC with ISH with HER2/CEP17 ratio ≥2).
6. Radiographically measurable disease according to RECIST 1.1 within 28 days prior to registration.
7. Adequate organ function as defined in the table below. All screening labs to be obtained within 28 days prior to registration.

   * Absolute Neutrophil Count ≥ 1.5 x 10^9/L
   * Hemoglobin (Hgb) ≥ 9 g/dL (may have been transfused)
   * Platelets ≥ 100 x 10^9/L OR ≥ 75 x 10^9/L for patients who received Cycle 1 of mFOLFOX6 +/- trastuzumab prior to registration
   * Calculated creatinine clearance1 ≥ 30 mL/min OR creatinine ≤ 1.5 × upper limit of normal (ULN)
   * Bilirubin ≤ 1.5 × upper limit of normal (ULN) (Subjects with Gilbert's syndrome may be enrolled despite a total bilirubin level >1.5 mg/dL, if their conjugated bilirubin is < 1.5× ULN)
   * Aspartate aminotransferase (AST) ≤ 2.5 × ULN OR ≤ 5x ULN in patients with known liver metastases
   * Alanine aminotransferase (ALT) ≤ 2.5 × ULN OR ≤ 5x ULN in patients with known liver metastases
8. Left ventricular ejection fraction (LVEF) ≥ 50% or above the lower limit of the institutional normal range, whichever is lower.
9. Females of childbearing potential must have a negative serum pregnancy test at screening. NOTE: Females are considered of child bearing potential unless they are surgically sterile (have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are naturally postmenopausal for at least 12 consecutive months.
10. Females of childbearing potential and males must be willing to abstain from heterosexual activity or to use 2 forms of effective methods of contraception from the time of informed consent until 210 days after treatment discontinuation. The two contraception methods can be comprised of two barrier methods, or a barrier method plus a hormonal method.
11. As determined by the enrolling physician or protocol designee, ability of the subject to understand and comply with study procedures for the entire length of the study.

Exclusion Criteria:

1. Previous systemic therapy for stage IV disease - EXCEPT that patient may have received one cycle of mFOLFOX6 +/- trastuzumab within the 4 weeks prior to registration.
2. Active infection requiring intravenous systemic therapy.
3. Pregnant or breastfeeding (NOTE: breast milk cannot be stored for future use while the mother is being treated on study).
4. Treatment with any investigational drug within 28 days prior to registration.
5. Prior immune checkpoint inhibitor therapy (i.e. anti-CTLA-4, anti-PD-L1, anti-PD-1), or HER2-directed therapy (including trastuzumab)
6. Evidence of interstitial lung disease or active, non-infectious pneumonitis
7. Untreated brain metastasis or brain metastasis treated within 4 weeks prior to enrollment.
8. Known additional malignancy that is active and/or progressive requiring treatment; exceptions include basal cell or squamous cell skin cancer, in situ cervical or bladder cancer, or other cancer for which the subject has been disease-free for at least five years.
9. Serious cardiovascular event within 6 months prior to study entry, including myocardial infarction, malignant hypertension, severe/unstable angina, symptomatic congestive heart failure (≥ New York Heart Association Classification Class II), cerebral vascular accident, transient ischemic attack, or serious cardiac arrhythmia requiring medication.
10. History of organ allograft or allogeneic stem cell transplantation
11. Active autoimmune disease requiring systemic treatment in the past 3 months (for example with disease modifying agents, corticosteroids, or immunosuppressive drugs).

    Exceptions Include:
    * Subjects with endocrine diseases stable on replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) or hormone suppression.
    * Subjects that require intermittent use of bronchodilators, local steroid injections, or inhaled or topical steroids
    * Subjects with vitiligo, psoriasis, Sjogren's syndrome, or resolved childhood asthma/atopy
12. Current use of immunosuppressive medication, EXCEPT for the following: a. intranasal, inhaled, topical steroids, or local steroid injection (e.g., intra-articular injection); b. Systemic corticosteroids at physiologic doses ≤ 10 mg/day of prednisone or equivalent; c. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication).
13. Known history of testing positive for HIV or known acquired immunodeficiency syndrome.
14. Known history of Hepatitis B virus (HBV) or hepatitis C virus (HCV) infection. Subjects with laboratory evidence of cleared HBV and HCV infection will be permitted.
15. Vaccination within 4 weeks of the first dose of avelumab and while on trials is prohibited except for administration of inactivated vaccines.
16. Known prior severe hypersensitivity to investigational product or any component in its formulations, including known severe hypersensitivity reactions to monoclonal antibodies (NCI CTCAE v5 Grade ≥ 3).
17. Persisting toxicity related to prior therapy (NCI CTCAE v5 Grade > 1); however, alopecia, sensory neuropathy Grade ≤ 2, or other Grade ≤ 2 not constituting a safety risk based on investigator's judgment are acceptable.
18. Other severe acute or chronic medical conditions including immune colitis, inflammatory bowel disease, immune pneumonitis, pulmonary fibrosis or psychiatric conditions including recent (within the past year) or active suicidal ideation or behavior; or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with informed consent, the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-01-24 (Actual); Primary Completion 2020-09-11 (Actual); Study Completion 2022-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ashwin Somasundaram, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (7):
- United States (7):
  - City of Hope, Duarte, California
  - Winship Cancer Insititute of Emory University, Atlanta, Georgia
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - University of Iowa Hospital and Clinics, Iowa City, Iowa
  - Atlantic Health System, Morristown, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee MS, Chao J, Mulcahy MF, Kasi PM, Alistar AT, Mukherjee S, Akce M, Moore DT, McRee AJ, Somasundaram A. Phase II study of avelumab and trastuzumab with FOLFOX chemotherapy in previously untreated HER2-amplified metastatic gastroesophageal adenocarcinoma. Oncologist. 2025 Jul 4;30(7):oyaf195. doi: 10.1093/oncolo/oyaf195. PMID 40571483

RESULTS

PARTICIPANT FLOW:
Groups:
- Induction and Maintenance: Cycles 1-9; Induction; Cycle = 14 days
  mFOLFOX6
  * oxaliplatin 85 mg/m2 IV Day 1 and
  * leucovorin 400 mg/m2 IV Day 1 and
  * 5 fluorouracil 400 mg/m2 IV bolus and 2400 mg/m2 IV over 46 hours Day 1 and
  Trastuzumab 6 mg/kg IV loading dose C1D1 then Trastuzumab 4 mg/kg IV Day 1 and
  Avelumab 800 mg IV Day 1
  Cycles 10 and subsequent; Maintenance; Cycle = 14 days
  Trastuzumab 4 mg/kg Day 1 and Avelumab 800 mg Day 1
  Oxaliplatin: Oxaliplatin 85 mg/m2
  Leucovorin: Leucovorin 400 mg/m2
  5 fluorouracil: 5 fluorouracil 400 mg/m2 bolus and 2400 mg/m2 continuous infusion
  Trastuzumab: Trastuzumab 6 mg/kg loading dose C1D1 then 4 mg/kg Day 1
  Avelumab: Avelumab 800 mg
Period: Overall Study
Arm/Group | Induction and Maintenance
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Induction and Maintenance
Number analyzed (Participants) | 18
Age, Continuous [Median (Full Range); unit: years] | 63 [46 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 18
Primary Tumor Site [Count of Participants; unit: Participants]
  Esophagus | 4
  Gastroesophageal Junction | 8
  Stomach | 4
  Not described or multiple | 2
HER2 IHC [Count of Participants; unit: Participants] — The IHC (immunohistochemistry) test gives a score of 0 to 3+ that measures the amount of HER2 (human epidermal growth factor receptor 2) receptor protein on the surface of cells in a breast cancer tissue sample. If the score is 0 to 1+, it's called HER2 negative. If the score is 2+, it's called borderline. A score of 3+ is called HER2 positive.
  Participants
    3 + | 12
    2+ with ISH (in situ hybridization) + | 6
Programmed cell death ligand 1(PD-L1) CPS Score [Count of Participants; unit: Participants] — Combined positive score (CPS) is defined as the number of positive tumor cells, lymphocytes and macrophages, divided by the total number of viable tumor cells multiplied by 100. A lower CPS score means better outcome or less positive cells.
  Participants
    CPS = 0 | 4
    CPS = 1 to <5 | 5
    CPS = 5 to <10 | 4
    CPS ≥ 10 | 4
    Unknown | 1

OUTCOME MEASURES:

1. Primary Outcome: Best Objective Response Rate (bORR)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST): Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter(LD) of target lesions; Progressive Disease (PD): >= 20% increase in tumor burden relative to nadir or the appearance of one or more new lesions; Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started.
  The bORR will be defined as the percentage of subjects whose best response by 24 weeks are either a CR or PR according to RECIST 1.1. For confirmed response, PR or CR need to be confirmed by repeat assessments that should be performed no less than 4 weeks. Otherwise, it will be considered as an unconfirmed response.
Time Frame: 24 weeks
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Induction and Maintenance
Number analyzed (Participants) | 18
Percentage of participants
  Best response rate (confirmed or unconfirmed) | 61 [39 to 84]
  Best confirmed response rate | 50 [29 to 71]

2. Secondary Outcome: Progression Free Survival (PFS)
Description: Per RECIST 1.1: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter(LD) of target lesions; Progressive Disease (PD): >= 20% increase in tumor burden relative to nadir or the appearance of one or more new lesions; Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started.
  Progression Free Survival (PFS) will be defined as the time from the start date of treatment to the date of documented progression as determined by RECIST 1.1 or death from any cause.
Time Frame: Time of treatment start until the criteria for disease progression or death, up to a maximum of 11 months.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Induction and Maintenance
Number analyzed (Participants) | 18
months | 8 [5.3 to NA] — The upper limit could not be reached due to insufficient number of participants with events.

3. Secondary Outcome: Progression Free Survival by iRECIST(iPFS)
Description: Immune-RECIST Criteria(iRECIST): Complete Response(iCR), Disappearance of all measurable and non-measurable lesions; Partial Response (iPR), >=30% decrease in tumor burden relative to baseline; Unconfirmed Progressive Disease (iUPD), >= 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions; Confirmed Progressive Disease (iCPD), confirmation of iUPD (by further growth) at the next assessment; Stable Disease (iSD), neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started.
  iPFS will be defined as the time from the start date of treatment to the date of documented progression as determined by iRECIST criteria or death from any cause.
Time Frame: Time of treatment start until the criteria for disease progression or death, up to a maximum of 11 months.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Induction and Maintenance
Number analyzed (Participants) | 18
months | 8 [5.3 to NA] — The upper limit could not be reached due to the insufficient number of participants with events.

4. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival (OS) will be defined as the time from start of treatment to the date of death from any cause, or date of last contact (censored).
Time Frame: Time of treatment start until death or date of last contact, up to a maximum of 20 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Induction and Maintenance
Number analyzed (Participants) | 18
months | 13.1 [11.5 to NA] — The upper limit could not be reached due to the insufficient number of participants with events.

5. Secondary Outcome: Disease Control Rate (DCR)
Description: Disease Control Rate (DCR) will be defined as the total number of patients whose best responses are either a CR, PR, or SD divided by the number of response evaluable patients. Patients with best response of SD will need to maintain SD by 24 weeks to be considered to have received clinical benefit from the treatment regimen.
Time Frame: Up to a maximum of 11 months.
Measure: Number; unit: Percentage of participants
Arm/Group | Induction and Maintenance
Number analyzed (Participants) | 18
Percentage of participants | 55.6

6. Secondary Outcome: Number of Participants With Grade 3-4 Treatment Related Adverse Events
Description: The frequency and severity of all grade 3-4 treatment related adverse events are reported by CTCAE v5.
Time Frame: AE had been recorded from time of signed informed consent until 30 days after discontinuation of study drug(s) and/or until a new anti-cancer treatment starts, whichever occurs first, up to a maximum of 20 months.
Measure: Number; unit: Participants
Arm/Group | Induction and Maintenance
Number analyzed (Participants) | 18
Participants
  Neutrophil count decreased | 6
  Platelet count decreased | 2
  Anemia | 2
  White blood cell decreased | 1
  Lymphocyte count decreased | 1
  Hypokalemia | 2
  Diarrhea | 2
  Gastroesophageal reflux disease | 1
  Lung infection | 1
  Mucositis oral | 1

ADVERSE EVENTS:
Time Frame: Up to a maximum of 20 months.
Arm/Group | Induction and Maintenance
All-Cause Mortality (participants affected / at risk) | 9/18
Serious Adverse Events (participants affected / at risk) | 7/18
Other Adverse Events (participants affected / at risk) | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Induction and Maintenance (N=18)
CARDIAC ARREST (Cardiac disorders) | 1 (1)
DIZZINESS (Nervous system disorders) | 1 (3)
FALL (Injury, poisoning and procedural complications) | 1 (2)
HEMATOMA (Vascular disorders) | 1 (1)
LUNG INFECTION (Infections and infestations) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 1 (2)
OBSTRUCTION GASTRIC (Gastrointestinal disorders) | 1 (3)
PLATELET COUNT DECREASED (Investigations) | 1 (2)
SEPSIS (Infections and infestations) | 1 (1)
THROMBOEMBOLIC EVENT (Vascular disorders) | 1 (2)
TUMOR HEMORRHAGE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
VOMITING (Gastrointestinal disorders) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Induction and Maintenance (N=18)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 2 (2)
ABDOMINAL PAIN (Gastrointestinal disorders) | 5 (8)
AGITATION (Psychiatric disorders) | 1 (1)
ALKALINE PHOSPHATASE INCREASED (Investigations) | 6 (10)
ALLERGIC RHINITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
ANEMIA (Blood and lymphatic system disorders) | 11 (35)
ANOREXIA (Metabolism and nutrition disorders) | 9 (13)
ANXIETY (Psychiatric disorders) | 2 (3)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 3 (6)
ASCITES (Gastrointestinal disorders) | 1 (1)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 3 (8)
BELCHING (Gastrointestinal disorders) | 2 (2)
BLOOD AND LYMPHATIC SYSTEM DISORDERS - OTHER, SPECIFY (Blood and lymphatic system disorders) | 1 (2)
BLOOD BILIRUBIN INCREASED (Investigations) | 3 (5)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 2 (2)
BRUISING (Injury, poisoning and procedural complications) | 2 (2)
CARDIAC DISORDERS - OTHER, SPECIFY (Cardiac disorders) | 2 (6)
CHILLS (General disorders) | 4 (4)
COLITIS (Gastrointestinal disorders) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 8 (10)
COUGH (Respiratory, thoracic and mediastinal disorders) | 5 (5)
CREATININE INCREASED (Investigations) | 4 (4)
DEHYDRATION (Metabolism and nutrition disorders) | 3 (3)
DEPRESSION (Psychiatric disorders) | 1 (1)
DIARRHEA (Gastrointestinal disorders) | 8 (25)
DIZZINESS (Nervous system disorders) | 4 (5)
DRY MOUTH (Gastrointestinal disorders) | 1 (1)
DYSESTHESIA (Nervous system disorders) | 1 (1)
DYSGEUSIA (Nervous system disorders) | 6 (10)
DYSPHAGIA (Gastrointestinal disorders) | 3 (11)
DYSPHASIA (Nervous system disorders) | 1 (1)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 2 (2)
EDEMA FACE (General disorders) | 1 (1)
EDEMA LIMBS (General disorders) | 4 (7)
EJECTION FRACTION DECREASED (Investigations) | 1 (1)
ENCEPHALOPATHY (Nervous system disorders) | 1 (2)
EOSINOPHILIA (Blood and lymphatic system disorders) | 1 (1)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 2 (3)
ESOPHAGEAL PAIN (Gastrointestinal disorders) | 2 (2)
FALL (Injury, poisoning and procedural complications) | 1 (1)
FATIGUE (General disorders) | 11 (18)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1)
FEVER (General disorders) | 2 (3)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 1 (2)
FLATULENCE (Gastrointestinal disorders) | 2 (2)
GAIT DISTURBANCE (General disorders) | 2 (2)
GASTROESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 3 (7)
GASTROINTESTINAL DISORDERS - OTHER, SPECIFY (Gastrointestinal disorders) | 4 (5)
GASTROINTESTINAL PAIN (Gastrointestinal disorders) | 2 (2)
GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS - OTHER, SPECIFY (General disorders) | 3 (3)
GENERALIZED MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 2 (3)
HEADACHE (Nervous system disorders) | 2 (2)
HEARING IMPAIRED (Ear and labyrinth disorders) | 1 (1)
HEMATOMA (Vascular disorders) | 1 (1)
HEMOLYTIC UREMIC SYNDROME (Blood and lymphatic system disorders) | 1 (1)
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 2 (2)
HOT FLASHES (Vascular disorders) | 1 (1)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 1 (2)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 2 (2)
HYPERKALEMIA (Metabolism and nutrition disorders) | 1 (2)
HYPERTENSION (Vascular disorders) | 7 (90)
HYPERTHYROIDISM (Endocrine disorders) | 1 (1)
HYPOALBUMINEMIA (Metabolism and nutrition disorders) | 6 (20)
HYPOCALCEMIA (Metabolism and nutrition disorders) | 2 (2)
HYPOGLYCEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPOKALEMIA (Metabolism and nutrition disorders) | 5 (10)
HYPOMAGNESEMIA (Metabolism and nutrition disorders) | 5 (10)
HYPONATREMIA (Metabolism and nutrition disorders) | 5 (10)
HYPOPHOSPHATEMIA (Metabolism and nutrition disorders) | 3 (8)
HYPOTENSION (Vascular disorders) | 2 (3)
HYPOTHERMIA (General disorders) | 1 (1)
HYPOTHYROIDISM (Endocrine disorders) | 1 (1)
INFECTIONS AND INFESTATIONS - OTHER, SPECIFY (Infections and infestations) | 2 (3)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 4 (9)
INJURY, POISONING AND PROCEDURAL COMPLICATIONS - OTHER, SPECIFY (Injury, poisoning and procedural complications) | 3 (4)
INSOMNIA (Psychiatric disorders) | 2 (2)
INVESTIGATIONS - OTHER, SPECIFY (Investigations) | 2 (3)
LOCALIZED EDEMA (General disorders) | 1 (1)
LYMPHOCYTE COUNT DECREASED (Investigations) | 5 (14)
MALAISE (General disorders) | 1 (2)
MUCOSITIS ORAL (Gastrointestinal disorders) | 4 (7)
MUSCLE WEAKNESS LOWER LIMB (Musculoskeletal and connective tissue disorders) | 2 (2)
MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDER - OTHER, SPECIFY (Musculoskeletal and connective tissue disorders) | 3 (3)
NAIL CHANGES (Skin and subcutaneous tissue disorders) | 1 (1)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 9 (18)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 2 (2)
NERVOUS SYSTEM DISORDERS - OTHER, SPECIFY (Nervous system disorders) | 1 (1)
NEUTROPHIL COUNT DECREASED (Investigations) | 11 (27)
NON-CARDIAC CHEST PAIN (General disorders) | 1 (4)
ORAL PAIN (Gastrointestinal disorders) | 1 (4)
PAIN (General disorders) | 1 (1)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 2 (3)
PALMAR-PLANTAR ERYTHRODYSESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 1 (1)
PALPITATIONS (Cardiac disorders) | 1 (1)
PARESTHESIA (Nervous system disorders) | 3 (7)
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 2 (2)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 12 (21)
PLATELET COUNT DECREASED (Investigations) | 9 (16)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 (2)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1 (2)
PRESYNCOPE (Nervous system disorders) | 1 (1)
PRURITUS (Skin and subcutaneous tissue disorders) | 3 (3)
RASH ACNEIFORM (Skin and subcutaneous tissue disorders) | 1 (1)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 4 (5)
RENAL AND URINARY DISORDERS - OTHER, SPECIFY (Renal and urinary disorders) | 2 (3)
RENAL CALCULI (Renal and urinary disorders) | 1 (1)
RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS - OTHER, SPECIFY (Respiratory, thoracic and mediastinal disorders) | 1 (1)
RHINORRHEA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
SEIZURE (Nervous system disorders) | 1 (1)
SINUS BRADYCARDIA (Cardiac disorders) | 1 (7)
SINUS TACHYCARDIA (Cardiac disorders) | 3 (4)
SKIN AND SUBCUTANEOUS TISSUE DISORDERS - OTHER, SPECIFY (Skin and subcutaneous tissue disorders) | 3 (5)
SORE THROAT (Respiratory, thoracic and mediastinal disorders) | 1 (1)
STOMACH PAIN (Gastrointestinal disorders) | 1 (1)
THYROID STIMULATING HORMONE INCREASED (Investigations) | 2 (2)
TINNITUS (Ear and labyrinth disorders) | 1 (1)
TUMOR HEMORRHAGE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
URINARY RETENTION (Renal and urinary disorders) | 3 (4)
URINARY TRACT INFECTION (Infections and infestations) | 1 (2)
UROSTOMY OBSTRUCTION (Injury, poisoning and procedural complications) | 1 (1)
VOMITING (Gastrointestinal disorders) | 7 (12)
WEIGHT GAIN (Investigations) | 1 (2)
WEIGHT LOSS (Investigations) | 8 (16)
WHITE BLOOD CELL DECREASED (Investigations) | 6 (29)
WOUND COMPLICATION (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-29): https://cdn.clinicaltrials.gov/large-docs/36/NCT03783936/Prot_SAP_000.pdf